CLINICAL TRIAL: NCT02737683
Title: Heterogeneous Distribution of Health Literacy and Emotional State on Patients With Functional Dyspepsia.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-Shun Wu, Director of GI / Visiting Staff, Taipei Medical University WanFang Hospital
Other Study IDs: N201601022
Record Dates: First submitted 2016-03-17; First posted 2016-04-14 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Dyspepsia
Keywords: Disease; anxiety; depression; combine; negative emotional states; functional dyspepsia
MeSH Terms: conditions — Dyspepsia; Disease; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with indigestion were often found in gastroenterology clinic, those who about 20 % was caused by organic, while the rest of patients are showed abnormal inspection, and these are so called functional dyspepsia. Functional dyspepsia is a chronic and repeated occurrence of digestive disorders, patients often visit hospitals frequently and unable to get fully cured. Current Symptom diagnoses are based on Rome III criteria as diagnostic criteria. Although functional dyspepsia condition should combine with physical and mental treatments, due to the reasons behind the complex, there is still no effective classification could be acted in health education and drug intervention.

DETAILED DESCRIPTION:
Health literacy can be defined as "ability for obtaining basic health information and understanding medical services." Within 10 years, healthy development and application of knowledge used in medical care and public health fields that have raised more attentions, many European countries set health knowledge as one of the main indicators for health care policy in the future. To promote behavior of self-care health for people, enhance the effective use of medical service , also reduce health care cost and unequally medical information.

Anxiety and depression are two common reactions when it comes to negative emotional states, which related to a body and caused a vicious cycle of disease. Some patients suffer from functional dyspepsia symptoms were diagnosed with anxiety or depression symptoms often ignore body care due to lack of health literacy. The purpose of this study is to investigate the distribution of functional dyspepsia patients with health literacy and emotional status, in order to provide more effective health education mode, thereby reducing the waste of medical resources, and promote patient health.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with functional dyspepsia , can Self-reading and the self-administered questionnaire.

Exclusion Criteria:

* Due to physical illness, cognitive ability is limited and other factors can not were completed self-administered questionnaires.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with functional dyspepsia , can Self-reading and the self-administered questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-01 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Symptom diagnoses are based on Rome III criteria as diagnostic criteria | up to 10 months to collect data and perform an analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shun Wu, Dr, Study Chair — Taipei Medical University WanFang Hospital
Locations (1):
- WanFangH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No